CLINICAL TRIAL: NCT07023718
Title: Study of a Cohort of 100 Patients on the Impact of Pelvic Joint Stiffness on the Fear of Falling in Subjects Aged Over 75 Years, Hospitalized or in Institution
Brief Title: Impact of Pelvic Joint Stiffness on the Fear of Falling in Subjects Aged Over 75 Years
Acronym: RAAPC
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Sud Ile-de-France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A01885-36
Record Dates: First submitted 2023-09-12; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2024-09

CONDITIONS: Fear of Falling; Pelvic Joint/Ligament Damage
Keywords: pelvic joint;; fear of falling; ankylosis
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The pelvic girdle is the mechanical structure at the center of the balance and walking systems. The lack of amplitude of the joints that compose it could induce a fear of falling, common in the geriatric population and often underdiagnosed with poorly identified risk factors. This study seeks to highlight an association between fear of falling and lack of amplitude of the different joints of the pelvic girdle in order to identify predisposed patients and to set up preventive measures and better medical care.

DETAILED DESCRIPTION:
The pelvic girdle is the mechanical structure at the center of the balance and walking systems. The lack of amplitude of the joints that compose it could induce a fear of falling, common in the geriatric population and often underdiagnosed with poorly identified risk factors. Fear of falling is defined as the enduring preoccupation with falling, leading the person to avoid activities that they are capable of doing. It modifies its behavior and affects its quality of life, its well-being and increases the risk of developing pathologies linked to the lack of physical activities. Joint stiffness is a major disorder in the elderly linked to bone and joint aging, but also to lack of mobilization. The pelvic girdle is the mechanical structure at the center of the balance and gait systems. The lack of amplitude of the joints that compose it could induce a fear of falling.

This study seeks to highlight whether there is an association between the fear of falling and the lack of amplitude of the different joints of the pelvic girdle.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged over 75 years hospitalized or in institution in the geriatric department of GHSIF (Groupe Hospitalier Sud -Ile-de France)

Exclusion Criteria:

* Patients that have undergone a lumbar surgery
* Patients with hospital diagnosed cognitive troubles

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Male and Female Subjects aged over 75 years old being hospitalized or in institution.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Association between fear of falling and articular stiffness | At inclusion
  The primary outcome is the association between joint stiffness and fear of falling:
  * Fear of falling assessed by FES-I (score).
  * Joint mobility assessed by Schober goniometry (degrees).
  * Joint mobility assessed by Schober index (centimeters).

SECONDARY OUTCOMES:
Validity of 3 FES-I categories based on anthropometric measurements | At inclusion
  Using the Falls Efficacy Scale - International (FES-I) questionnaire. It is an improved version of the Fall Efficacy Scale (FES) proposed by Tinetti (18). The FES-I was developed by the Prevention of Falls Network Europe (ProFaNE) group. It is available on the ProFaNE website. The scale includes 16 items, each scored from 1 (not at all concerned) to 4 (very concerned), resulting in a total score range from 16 to 64.
  FES-I scores are typically categorized as follows:
  Low concern: 16-19
  Moderate concern: 20-27
  High concern: 28-64
  Higher scores indicate a worse outcome, reflecting a greater fear of falling and decreased confidence in performing daily activities safely.

CONTACTS AND LOCATIONS:
Overall Officials: sylvie Aufaure, MD, Principal Investigator — Groupe Hospitalier Sud Ile-de-France
Locations (2):
- France (2):
  - EHPAD Brie Comte Robert, Brie-Comte-Robert, Île-de-France Region
  - Centre Hospitalier Melun, Melun, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT07023718/Prot_SAP_000.pdf